CLINICAL TRIAL: NCT07177950
Title: A Two-cohort Study of SHR-A1811 in the Treatment of HER2-positive Breast Cancer With Brain Metastases, With or Without Leptomeningeal Metastases.
Brief Title: A Two-cohort Study of SHR-A1811 in the Treatment of HER2-positive Breast Cancer With Brain Metastases
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-113
Record Dates: First submitted 2025-09-02; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Brain Metastases; Leptomeningeal Metastasis
Keywords: HER2-positive breast cancer; SHR-A1811
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms; Meningeal Carcinomatosis | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Systemic SHR-A1811 therapy combined with intrathecal SHR-A1811 therapy
  Interventions: Drug: SHR-A1811
- Arm 2 (Experimental): Systemic SHR-A1811 therapy combined with radiotherapy
  Interventions: Drug: SHR-A1811; Radiation: radiotherapy

INTERVENTIONS:
Drug: SHR-A1811 — Systemic therapy: 4.8 mg/kg administered as an intravenous infusion on Day 1 of each cycle. 3 weeks a cycle. Continuous medication until study completion, occurrence of intolerable toxicity, disease progression, withdrawal from the study for any reason, or death, whichever occurs first, or until the investigator deems that the patient would no longer benefit from the treatment.
Drug: SHR-A1811 — Intrathecal therapy: Administered intrathecally on Day 1 of each cycle. Dose escalation follows a Bayesian Optimal Interval (BOIN) design with three predefined dose levels-15 mg, 30 mg, and 40 mg. The starting dose level is 15 mg. Patients are enrolled in cohorts of three per dose level. If no dose-limiting toxicities (DLTs) are observed, escalation proceeds to the next higher dose level according to the BOIN algorithm. Treatment is administered for a minimum of two cycles and is continued until cerebrospinal fluid (CSF) cytology achieves negative conversion, completion of six cycles, or intolerable adverse events, whichever occurs first. Extension beyond six cycles may be permitted following investigator's discussion and must be documented with justification.
  Arms: Arm 1
Radiation: radiotherapy — radiotherapy is determined by investigator's choice
  Arms: Arm 2

SUMMARY:
This is a multi-center, open-label, two-cohort study. The purpose of this study is to evaluate the safety, tolerability and efficacy of SHR-A1811 in the treatment of HER2-positive breast cancer with brain and leptomeningeal metastases, and the efficacy and safety of SHR-A1811 in the treatment of HER2-positive breast cancer with brain but without leptomeningeal metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-75 years (inclusive).
2. Histologically or cytologically confirmed HER2-positive advanced breast cancer (IHC 3+, or IHC 2+ with ISH amplification).
3. Radiologically documented brain metastases, with or without baseline leptomeningeal disease:

   * Cohort A (leptomeningeal metastasis cohort): leptomeningeal involvement demonstrated by contrast-enhanced MRI or positive cerebrospinal fluid (CSF) cytology.
   * Cohort B (no leptomeningeal metastasis cohort): ≥1 measurable intracranial lesion; either CNS-naïve or progressive after prior local therapy.
4. Anticipated life expectancy >12 weeks.
5. ECOG performance status 0-2.
6. Adequate organ function as defined by the following laboratory criteria:

   1. Hematologic: absolute neutrophil count (ANC) ≥1.5 × 10⁹/L, platelet count (PLT) ≥100 × 10⁹/L, hemoglobin (HGB) ≥90 g/L.
   2. Hepatic: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × upper limit of normal (ULN) (≤5 × ULN in patients with liver metastases); total serum bilirubin (TBIL) ≤1.5 × ULN; serum albumin ≥30 g/L.
   3. Renal: serum creatinine (Cr) ≤1.5 × ULN or calculated creatinine clearance ≥50 mL/min using the Cockcroft-Gault formula.
   4. Coagulation: prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤1.5 × ULN.
   5. Cardiac: left ventricular ejection fraction (LVEF) ≥50%.
7. Negative serum pregnancy test; women of childbearing potential must use a highly effective contraceptive method from study initiation until at least 6 months after the last dose of study medication.
8. Voluntary participation with written informed consent obtained prior to any study-related procedures.

Exclusion Criteria:

1. Cohort A participants must be excluded if any of the following apply:

   1. Cerebrospinal fluid (CSF) circulation obstruction that cannot be adequately controlled by therapeutic measures.
   2. MRI evidence of nodular leptomeningeal (LM) disease in the setting of negative CSF cytology.
   3. Active central nervous system (CNS) infection.
   4. Clinically significant coagulopathy.
2. Cohort B participants must be excluded if leptomeningeal metastasis is documented, defined as either: radiographic evidence of leptomeningeal involvement, or positive CSF cytology, or unequivocal clinical signs or symptoms attributable to leptomeningeal disease.
3. Presence of clinically significant third-space fluid accumulation (e.g., massive pleural or peritoneal effusion) that cannot be adequately controlled by drainage or other interventions.
4. Known hypersensitivity to any study drug or its excipients, or to any prior humanized monoclonal antibody products (e.g., trastuzumab, pertuzumab).
5. Prior or current exposure to antibody-drug conjugates (ADCs) containing a topoisomerase I inhibitor, including but not limited to fam-trastuzumab deruxtecan (DS-8201a).
6. Clinically significant cardiovascular disease, including but not limited to: severe or unstable angina pectoris, symptomatic congestive heart failure (New York Heart Association class ≥ II), clinically relevant supraventricular or ventricular arrhythmias requiring therapy or intervention, myocardial infarction within 6 months prior to first study dose, or cerebrovascular accident (including transient ischemic attack).
7. Participants known or suspected to interstitial lung disease.
8. Concurrent participation in any other interventional drug clinical trial.
9. Refusal to comply with protocol-mandated follow-up.
10. Presence of any additional severe physical or psychiatric disorder, or any laboratory abnormality that, in the investigator's judgment, could increase the subject's risk, confound study results, or render the patient unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 51 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
1. Number of Dose-Limiting Toxicities (DLTs) in the Sequential Dose-Escalation Cohort | Start of treatment until 3-week follow-up
  For cohort A. DLT is defined as any of the following events judged by the investigator to be related or possibly related to SHR-A1811 occurring within Cycle 1 (21 days), graded according to NCI-CTCAE v5.0:
  1. Grade ≥3 neurologic toxicity;
  2. Any death unless unequivocally attributable to tumor progression or an unrelated exogenous cause.
CNS-PFS | Start of treatment until 2-year follow-up
  For cohort B: Central nervous system- progression free survival: time from the date when the subject first received SHR-A1811 to the first observation of tumor progression of central nervous system or death from any cause.

SECONDARY OUTCOMES:
CNS-PFS | Start of treatment until 2-year follow-up
  For cohort A: Central nervous system- progression free survival: time from the date when the subject first received SHR-A1811 to the first observation of tumor progression of central nervous system or death from any cause.
CNS-ORR | Start of treatment until 2-year follow-up
  For cohort B. Central nervous system- objective response rate: proportion of subjects who achieved complete remission (CR) or partial remission (PR) of central nervous system by primary tumor imaging evaluation.
PFS | Start of treatment until 2-year follow-up
  Progression free survival: time from the date when the subject first received SHR-A1811 to the first observation of tumor progression or death from any cause.
OS | Start of treatment until 2-year follow-up
  Overall survival: time from the date when the subject first received SHR-A1811 to death from any cause.
Quality of life score | Start of treatment until 2-year follow-up
  Evaluated by the quality of life core scale [EORTC QLQ-C30 (Chinese version)] developed by European cancer research and treatment organization. The scope of each domain is 0 to 100. Higher scores in the functional and general health areas indicate better functional status and quality of life, and higher scores in the symptomatic areas indicate more symptoms or problems (poorer quality of life).
Incidence and severity of adverse events (AE) and serious adverse events (SAE) | Start of treatment until 2-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bin Shao, Principal Investigator — Peking University Cancer Hospital & Institute; Xiaoyan Li, Principal Investigator — Beijing Tiantan Hospital

IPD SHARING:
Plan to Share IPD: No